CLINICAL TRIAL: NCT00157963
Title: A 12 Week, Open, Randomized, Parallel, Multicenter Study of Efficacy, Tolerability & Safety of Hydrochlorothiazide (+) Losartan Potassium Versus Amlodipine in Essential Hypertensive Patients.
Brief Title: Hydrochlorothiazide (+) Losartan Potassium vs. Amlodipine Comparative Study (0954A-314)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-314; 2005_067
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Hydrochlorothiazide; Losartan; Duration of Therapy

INTERVENTIONS:
Drug: MK0954A; hydrochlorothiazide (+) losartan potassium / Duration of Treatment: 12 weeks

SUMMARY:
An efficacy and safety study of hydrochlorothiazide (+) losartan potassium compared to amlodipine at week 12 in Korean patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 20 70 75 with essential hypertension
* SiDBP 90 ~ 114mmHg at V1 & V2

Exclusion Criteria:

* Patient has known or suspected secondary hypertension
* Patient has a history of malignant hypertension (SiSBP > 210mmHg)
* Individuals has a known sensitivity or intolerance to HCTZ or any AIIAs, or any sulfonamide-derived drugs.
* Patient has shown significant abnormal laboratory evaluations

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2005-02-05 (Actual); Primary Completion 2006-02-08 (Actual); Study Completion 2006-02-08 (Actual)

PRIMARY OUTCOMES:
Antihypertensive efficacy of 12 weeks of treatment with hydrochlorothiazide (+) losartan potassium/amlodipine

SECONDARY OUTCOMES:
Safety/Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Chung JW, Lee HY, Kim CH, Seung IW, Shin YW, Jeong MH, Cho MC, Oh BH. Losartan/Hydrochlorothiazide fixed combination versus amlodipine monotherapy in korean patients with mild to moderate hypertension. Korean Circ J. 2009 Apr;39(4):151-6. doi: 10.4070/kcj.2009.39.4.151. Epub 2009 Apr 28. PMID 19949604